CLINICAL TRIAL: NCT05523154
Title: Nanopore Sequencing for Detecting Bacteria in Bile and Preventing Surgical Site Infections in Patients Undergoing Surgery for Benign or Malignant Pancreatic Tumors
Brief Title: "Answers in Hours" A Randomized Controlled Trial Using Microbiome Metagenomics for Bile Duct Cultures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-004234; NCI-2022-06735 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-08-23; First posted 2022-08-31 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Benign Pancreatic Neoplasm; Malignant Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Specimen Handling; Clinical Laboratory Techniques; Nanopore Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (biospecimen collection, routine testing) (Active Comparator): Patients undergo the collection of bile samples during standard of care surgery. Samples undergo routine laboratory testing.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Procedure
- Arm II (biospecimen, nanopore sequencing, routine testing) (Experimental): Patients undergo the collection of bile samples during standard of care surgery. Samples undergo nanopore sequencing and routine laboratory testing.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Procedure; Device: Nanopore Sequencing

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of bile samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Laboratory Procedure — Undergo routine laboratory testing
  Other Names: lab exam; Lab Test; Lab Tests; lab_exam; Laboratory Test; laboratory_test; Test; Tests
Device: Nanopore Sequencing — Undergo nanopore sequencing
  Other Names: Oxford Nanopore; Oxford Nanopore Sequencing; Oxford Nanopore Sequencing Technology
  Arms: Arm II (biospecimen, nanopore sequencing, routine testing)

SUMMARY:
This trial evaluates whether testing of bile with nanopore sequencing results in earlier detection of bacteriobilia (bacteria in bile) that may lead to surgical site infections in patients undergoing surgery for benign or malignant pancreatic tumors. Surgical site infections are a significant source of poor outcomes in patients undergoing surgery for pancreatic tumors. In most patients who develop this kind of infection, the bacteria identified as causing the infection is also frequently found to be in the bile at time of surgery. Usage of nanopore sequencing for detection of bacteria in the bile of patients undergoing surgery may allow doctors to prevent surgical site infections or treat them sooner or more effectively.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To improve antibiotic stewardship (reducing duration of peri-operative prophylactic antibiotic regimen, reducing administration of broad-spectrum antibiotic) by providing surgical team with rapid Oxford Nanopore (ONT) sequencing data in the early post-operative setting.

SECONDARY OBJECTIVE:

I. To reduce the cost of care through reduction in surgical site infection (SSI) and improved antibiotic stewardship.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo the collection of bile samples during standard of care surgery. Samples undergo routine laboratory testing.

ARM II: Patients undergo the collection of bile samples during standard of care surgery. Samples undergo nanopore sequencing and routine laboratory testing.

After completion of study, patients' medical records are reviewed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 year (yr) male (M) or female (F)
* Undergoing pancreaticoduodenectomy or total pancreatectomy for any benign or malignant indication with informed consent

Exclusion Criteria:

* Women who are pregnant
* Patients who are institutionalized or incarcerated
* Patients without the cognitive capacity to consent
* Patients undergoing emergency pancreaticoduodenectomy or total pancreatectomy
* Patients enrolled in similar clinical trials involving use of perioperative antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina R. Walther-Antonio, PhD, Principal Investigator — Mayo Clinic in Rochester; Mark J. Truty, MD, MS, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study evaluated the clinical use of Oxford Nanopore Sequencing in characterizing biliary microbial contamination in patients undergoing pancreatic head resection (total pancreatectomy, pancreaticoduodenectomy) surgery. Following enrollment, stratified randomization was performed using surgery type as a stratification factor. Patients that did not complete surgery were, therefore, removed from the study prior to assignment to a study group.
  assignment to a study group was dependent
Period: Overall Study
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing) | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (19.14) | 55.8 (15.32) | 56.5 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infections
Description: Assessed by incidence of surgical site infections (SSI), classified using American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) definitions. Diagnostics tests to evaluate for SSI included physical examination, laboratory testing, and imaging such as computed tomography (CT) and ultrasound (US). Patients with complicated hospital courses returned for clinical visit after approximately 2 weeks with cross sectional CT imaging and laboratory testing with further follow up visits as clinically indicated. In the instance of an uneventful hospital course, patients returned at 4 weeks from their date of discharge for a clinical visit with CT imaging and laboratory testing. After this first routine follow-up appointment with surgery, patients continued to follow with medical oncology and with the surgical clinic on an as needed basis.
Time Frame: Up to 90 days
Population: To determine whether the use of rapid Oxford Nanopore sequencing technology reduced rates of surgical site infections we compared the number of patients diagnosed with a surgical site infection in Arm II compared to the number of patients diagnosed with a surgical site infection in Arm I.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
Number analyzed (Participants) | 3 | 5
Participants | 1 | 2

2. Primary Outcome: Improved Antibiotic Stewardship - Number of Antibiotics
Description: Assessed by the total number of antibiotics administered.
Time Frame: Up to 90 days
Population: To determine whether use of Oxford Nanopore sequencing improved antibiotic stewardship we compared the total number of antibiotics administered to Arm II patients compared to the total number of antibiotics administered to Arm I patients. We also compared the number of days patients were on antibiotics
Measure: Mean (Standard Deviation); unit: Antibiotics Administered
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
Number analyzed (Participants) | 3 | 5
Antibiotics Administered | 7.7 (2.31) | 5.4 (1.82)

3. Primary Outcome: Improved Antibiotic Stewardship - Duration
Description: Assessed by the number of days patients were on antibiotics.
Time Frame: Up to 90 days
Population: To determine whether use of Oxford Nanopore sequencing improved antibiotic stewardship we compared the total number of days patients were on antibiotics to Arm II patients compared to the total number of days patients were on antibiotics to Arm I patients.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
Number analyzed (Participants) | 3 | 5
Days | 21 (14.93) | 25.2 (23.30)

4. Secondary Outcome: Timeliness of Sample Analysis
Description: Assessed by the time from sample collection to completion of sample analysis, reported in hours.
Time Frame: Up to 90 days
Population: To determine whether use of Oxford Nanopore Sequencing resulted in more rapid microbial results we compared the time taken to complete microbial standard cultures in Arm with the time taken to complete Oxford Nanopore sequencing analysis in Arm II.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
Number analyzed (Participants) | 3 | 5
Hours | 163.5 (87.56) | 60.9 (2.32)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 90 days post-surgery. Adverse events were assessed daily while inpatient and then weekly while outpatient
Description: All recorded adverse events are reported. These include all adverse events Grade III or higher (requiring surgical, endoscopic, or radiological intervention) and all observed or volunteered adverse effects Grade III or higher (serious or non-serious) and abnormal test findings, regardless of the treatment group if applicable or suspected causal relationship to the investigational device (Oxford Nanopore sequencing) or if applicable to other study treatment or diagnostic product(s).
Arm/Group | Arm I (Biospecimen Collection, Routine Testing) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Biospecimen Collection, Routine Testing) (N=3) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing) (N=5)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Intraabdominal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Bactereremia (Infections and infestations) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal infection/ bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Biospecimen Collection, Routine Testing) (N=3) | Arm II (Biospecimen, Nanopore Sequencing, Routine Testing) (N=5)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Nausea/ vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Post-operative biliary leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomal ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was limited in that it was terminated early resulting in a small number of subjects being analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05523154/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT05523154/ICF_001.pdf